CLINICAL TRIAL: NCT07267325
Title: The Effect of Exercise With or Without Antiresorptive Therapy, on Bone Properties in Postmenopausal Women With Low BMD - Randomised Controlled Unilateral Intervention Trial
Brief Title: Bone Health in Postmenopausal Women: The Effect of Exercise With or Without Medication for Osteoporosis
Acronym: BEAT-OP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Loughborough University (Other)
Collaborators: University of Sheffield (Other); University of Cambridge (Other)
Responsible Party: Principal Investigator, Katherine Brooke-Wavell, Professor, Loughborough University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 354429
Record Dates: First submitted 2025-11-14; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-10

CONDITIONS: Osteoporosis in Post-menopausal Women
Keywords: Exercise; Bone mineral density; Bone strength; Bone geometry; Fracture risk; Bone structure; Biomarkers
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The researcher conducting imaging assessments and analyses will remain blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Without any medication affecting bone (Experimental): Participants in this arm are postmenopausal women with low bone density who are not taking any bone medication for at least 12 months. They will participate in a 12-month supervised high impact unilateral hopping exercise.
  Interventions: Behavioral: EXERCISE TRAINING
- With osteoporosis medication (antiresorptive ) (Experimental): Participants in this arm are postmenopausal women with low bone density who are taking antiresorptive medication for at least 12 months. They will participate in a 12-month supervised high impact unilateral hopping exercise.
  Interventions: Behavioral: EXERCISE TRAINING; Drug: Antiresorptive medication (routine clinical care)

INTERVENTIONS:
Behavioral: EXERCISE TRAINING — The unilateral high-impact (hopping) exercise will be on one randomly allocated exercise leg, with the contralateral leg being untrained to provide a control leg. Each session will begin with a warm-up targeting the legs and lower back. The progressive exercise regimen consists of multidirectional hopping exercises that will gradually increase in technique, intensity, and frequency to ensure safety. It will be personalised according to the participants' physical abilities and responses during or after the exercise.
Drug: Antiresorptive medication (routine clinical care) — Participants in this arm are already taking prescribed antiresorptive medication as part of standard clinical care. The study will not provide or modify the medication.
  Arms: With osteoporosis medication (antiresorptive )

SUMMARY:
Osteoporosis is a systemic bone disorder characterised by a reduced bone mass and structural deterioration, increasing the risk of fragility fractures, particularly in women post-menopause. Bone mass and structure can be assessed by scans.

Antiresorptive medications are commonly prescribed to reduce bone resorption, preventing further bone loss and thus reducing the possibility of fracture. Exercise can also benefit bone mass and structure but current evidence do not show whether exercise is more, or less, effective in combination with antiresorptive medication.

This study will compare the effect of a brief, home-based exercise programme on bone mineral and structural properties in women taking/ not taking antiresorptive medication.

DETAILED DESCRIPTION:
Exercise can benefit bone density and induce structural changes, leading to a decrease in fracture risk. High-impact exercise is often recommended for promoting bone health as it generates the brief, high strains that stimulate bone adaptation. Brief multidirectional hopping exercises have been demonstrated to be a practical and sustainable intervention with older men, pre- and postmenopausal women. They allow exercise to be conducted on one leg, whilst changes in the other leg can be used as a control to compare what would happen without exercise.

The effects of exercise on bone density and structure may be different in women taking osteoporosis medication, but few studies have examined this group. This study thus aims to evaluate the effects of exercise on bone density and structure according to osteoporosis medication use.

The study will be a 12-month long randomised controlled trial including two groups: with and without antiresorptive osteoporosis medication for at least 12 months. Participants must not plan to change their treatment choices during the 12-month study. All participants will complete a 12-month unilateral hopping exercise intervention.

Screening and baseline measurements will include dual X-ray absorptiometry (DXA) and computed tomography (CT) scans of the hip, blood collection, hop assessment and questionnaires. Eligible participants will then be invited to commence the exercise intervention and randomly allocated an exercise leg, with the contralateral leg being untrained to provide a control leg. Randomisation of exercise and control legs will be performed by selecting an opaque sealed envelopes which contain "R" or "L" letters. It is not possible to blind the participant or researchers supervising the intervention to leg allocation.

An initial familiarisation session will be conducted under supervision. The exercise intervention involves a home-based exercise programme starting at three days per week, with the goal of increasing to seven days per week. It will begin with a warm-up targeting the legs and lower back, followed by a progressive exercise regimen that will gradually increase in technique, intensity, and frequency to ensure safety. It will be personalised according to the participants' physical abilities and responses during or after the exercise. Weekly supervised group sessions will be offered, and used to advise participants on progression of exercise. An exercise logbook will monitor adherence. A questionnaire on any injuries, soreness, or discomfort will be administered monthly online or by phone. Participants will be instructed to reduce intensity and frequency or discontinue exercise if they experience any adverse symptoms or discomfort.

Follow-up measurements will be conducted six and twelve months after the start of the exercise intervention is completed. All measurements , except for the CT scan, will also be repeated after six months with each visit expected to last no more than two hours. whereas at twelve months, all measurements will be repeated. CT scans will take place at Glenfield Hospital, Leicester. All other visits will take place at Loughborough University.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 55-75 years old
* >4y since menopause/hysterectomy/oophorectomy.
* Baseline femoral neck or lumber spine BMD T-score between -1 and -3.
* Able to complete the hopping exercises.
* Have no regular involvement for more than once/week in:

  1. Strength, powerlifting or high load resistance exercise.
  2. High to moderate impact exercise that known to involve ground reaction forces 2 to 4 times greater than body weight (e.g. Jogging).
* Treatment group: taking antiresorptive treatment for osteoporosis continuously for at least 12 months, and who intend to continue this medication for the rest of the study.
* Control group: not taking any medication affecting bone and no intention to commence such medication for the rest of the study.

Exclusion Criteria:

* Body mass index (BMI) >35 kg/m2
* Any medical condition, surgery, or injuries that contraindicate exercises including lower limb or back pain, knee or hip osteoarthritis.
* Vertebral fracture or multiple low trauma fractures (recent expert consensus recommends lower impact exercise for these groups)
* Replacement of hip joint(s)

Ages: 55 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Femoral neck bone mineral content BMC | Baseline, 6 months and 12 months
  (g) measured by DXA
Femoral neck bone mineral density BMD | Baseline, 6 months and 12 months
  (g/cm^2) measured by DXA

SECONDARY OUTCOMES:
Total hip bone mineral content BMC | Baseline, 6 months and 12 months
  (g) measured by DXA
Total hip bone mineral density BMD | Baseline, 6 months and 12 months
  (g/cm^2) measured by DXA
Lumbar spine bone mineral content BMC | Baseline, 6 months and 12 months
  (g) measured by DXA
Lumbar spine bone mineral density BMD | Baseline, 6 months and 12 months
  (g/cm^2) measured by DXA
Prevalent vertebral fracture | Baseline, 6 months and 12 months
  assessed using DXA vertebral morphology
Whole body composition | Baseline, 6 months and 12 months
  weight in Kg
Whole body composition | Baseline, 6 months and 12 months
  Hight in cm
Total fat mass | Baseline, 6 months and 12 months
  will be measured using whole body DXA, reported in Kg
Lean mass | Baseline, 6 months and 12 months
  will be measured using whole body DXA, reported in Kg
Tibia distal (4%) Total volumetric bone density vBMD | Baseline, 6 months and 12 months
  (mg/cm^3) measured by pQCT
Tibia distal (4%) trabecular density vBMD | Baseline, 6 months and 12 months
  (mg/cm^3) measured by pQCT
Tibia distal (4%)Total bone area | Baseline, 6 months and 12 months
  (mm) measured by pQCT
Tibia shaft (66%) cortical content per 1 mm | Baseline, 6 months and 12 months
  (mg/mm) measured by pQCT
Tibia shaft (66%) cortical thickness | Baseline, 6 months and 12 months
  (mm) measured by pQCT
Tibia shaft (66%) cortical vBMD | Baseline, 6 months and 12 months
  (mg/cm^3) measured by pQCT
Femoral neck integral BMC | Baseline and 12 months
  g measured by QCT
Femoral neck cortical BMC | Baseline and 12 months
  g measured by QCT
Femoral neck trabecular BMC | Baseline and 12 months
  g measured by QCT
Proximal femur cortical thickness | Baseline and 12 months
  mm measured by QCT
Plasma bone turnover biomarkers (resorption marker) | Baseline, 6 months and 12 months
  Bone turnover will be assessed using blood samples to measure C-terminal telopeptide of type I collagen (CTX) which will be reported in µg/L where higher values reflect higher bone turnover, which is associated with increased bone loss
Hop performance (ground reaction force). | Baseline, 6 months and 12 months
  measured by force plate reported in Newtons (N)
Total Bone-specific Physical Activity Questionnaire (BPAQ) score | Baseline and 12 months
  Total score from the Bone specific Physical Activity Questionnaire will be calculated based on physical activity, intensity and frequency The questionnaire does not have a fixed minimum or maximum score, and values depend on each participant's activity history.
  Higher scores indicate higher levels of bone loading physical activity. The contribution of this activity to skeletal adaptation.
Daily calcium intake | Baseline, 6 months and 12 months
  (mg) Calcium Questionnaire
Fall and balance confidence | Baseline, 6 months and 12 months
  will be assessed using Short Falls Efficacy Scale International (short- FES-I). The scale includes 7 items, each scored from 1 (Not at all concerned) to 4 (Very concerned).
  Total scores range from 7 to 28, where higher scores indicate lower confidence and greater fear of falling.
Trochanter BMD | Baseline, 6month and 12month
  g/cm^2 by DXA
Trochanter BMC | Baseline, 6month and 12month
  g by DXA
Tibia shaft (66%) cortical area | Baseline, 6 months and 12 months
  (mm^2) measured by pQCT
Tibia shaft (66%) Periosteal circumference | Baseline, 6 months and 12 months
  (mm) measured by pQCT
Tibia shaft (66%) Endosteal circumference | Baseline, 6 months and 12 months
  (mm) measured by pQCT
Tibia shaft (66%) Axial area moment of inertia | Baseline, 6 months and 12 months
  (mm^4) measured by pQCT
Tibia shaft (66%) Moment of resistance | Baseline, 6 months and 12 months
  (mm^3) measured by pQCT
Tibia shaft (66%) Total bone area | Baseline, 6 months and 12 months
  (mm^2) measured by pQCT
Tibia shaft (66%) Strength Strain Index | Baseline, 6 months and 12 months
  (mm^3) measured by pQCT
Trochanter integral BMC | Baseline and 12 months
  g measured by QCT
Trochanter cortical BMC | Baseline and 12 months
  g measured by QCT
Trochanter trabecular BMC | Baseline and 12 months
  g measured by QCT
Intertrochanter integral BMC | Baseline and 12 months
  g measured by QCT
Intertrochanter cortical BMC | Baseline and 12 months
  g measured by QCT
Intertrochanter trabecular BMC | Baseline and 12 months
  g measured by QCT
Mid-femoral neck geometry | Baseline and 12 months
  Buckling ratio measured by QCT
Mid-femoral neck geometry | Baseline and 12 months
  Cross-sectional moment of inertia minimum (cm^4) measured by QCT
Mid-femoral neck geometry | Baseline and 12 months
  Cross-sectional moment of inertia maximum (cm^4) measured by QCT
Mid-femoral neck geometry | Baseline and 12 months
  Cross-sectional moment of area (cm^2) measured by QCT

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Brooke-Wavell, Professor, Principal Investigator — Loughborough University
Locations (1):
- Loughborough University, Loughborough, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: No